CLINICAL TRIAL: NCT06367179
Title: Investigation of Learning Effectiveness and Self-efficacy of Caregivers in Pressure Injury Wound Care Before and After Virtual Reality and AI Wound-detecting System Intervention
Brief Title: Virtual Reality and AI Wound-detecting System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202401039RINC
Record Dates: First submitted 2024-03-24; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-02

CONDITIONS: Pressure Injury
Keywords: Virtual reality; wound care; Artificial Intelligence; Self-efficacy
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive interventions of virtual reality and artificial intelligence wound detecting system.
  Interventions: Other: Virtual reality and AI use
- Control group (Other): The control group maintained the traditional pressure injury health education with oral introduction and health education leaflet.
  Interventions: Other: Health education leaflet

INTERVENTIONS:
Other: Virtual reality and AI use — The experimental group will receive interventions of virtual reality and artificial intelligence wound detecting system.
  Arms: Experimental group
Other: Health education leaflet — The control group maintained the traditional pressure injury health education with oral introduction and health education leaflet.
  Arms: Control group

SUMMARY:
This study is an experimental study. The main caregivers of pressure injury patients in the plastics surgery ward and general medicine ward of the hospital in Taipei City who are over 20 years old, have good communication skills in Chinese and Taiwanese or who can read Chinese are the research objects. During the study process, pre-tests will be given to the accepted subjects, which are the correctness evaluation scale of caregiver's pressure injury wound dressing change and caregiver self-efficacy scale, and then the accepted subjects will be divided into experimental group and control group. The experimental group will receive interventions of virtual reality and artificial intelligence wound detecting system, while the control group maintained the traditional pressure injury health education with oral introduction and health education leaflet. After the intervention measures are given, a post-test (same as the pre-test content) will be conducted within two days. Finally, analyze the effectiveness of the intervention of virtual reality pressure injury education video and artificial intelligence wound detecting system on caregivers of pressure injury improve wound care correctness and increase self-efficacy.

DETAILED DESCRIPTION:
Pressure injury care is a great burden for caregivers from non-medical backgrounds. Due to low self-efficacy, caregivers often do not have enough confidence to perform correct wound dressing procedures, which leads to ineffective care of pressure wounds and causes the pressure injury patient's wound repeatedly inflamed and deteriorated. Therefore, the purpose of this study is to investigate the effectiveness of the intervention on the correctness of dressing change and self-efficacy of pressure injury caregivers through virtual reality of pressure injury education videos and artificial intelligence wound detecting system. This study is an experimental study. The main caregivers of pressure injury patients in the plastics surgery ward and general medicine ward of the hospital in Taipei City who are over 20 years old, have good communication skills in Chinese and Taiwanese or who can read Chinese are the research objects. During the study process, pre-tests will be given to the accepted subjects, which are the correctness evaluation scale of caregiver's pressure injury wound dressing change and caregiver self-efficacy scale, and then the accepted subjects will be divided into experimental group and control group. The experimental group will receive interventions of virtual reality and artificial intelligence wound detecting system, while the control group maintained the traditional pressure injury health education with oral introduction and health education leaflet. After the intervention measures are given, a post-test (same as the pre-test content) will be conducted within two days. Finally, analyze the effectiveness of the intervention of virtual reality pressure injury education video and artificial intelligence wound detecting system on caregivers of pressure injury improve wound care correctness and increase self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Actual age is over 20 years old.
2. Those who can communicate smoothly in Mandarin and Taiwanese, or those who have the ability to read Chinese.
3. Caregivers of patients with pressure injuries.

Exclusion Criteria:

1. Those who suffer from mental or intelligence-related diseases or whose cognitive abilities are insufficient to answer the questionnaire questions.
2. Those who are unable to complete basic demographic information.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-02-04 (Estimated); Study Completion 2025-02-04 (Estimated)

PRIMARY OUTCOMES:
Accurate dressing change rate of pressure injury | 2 days
  This scale mainly evaluates the correctness of dressing changes for pressure injuries. Three pressure injury scales are designed for stage 2 pressure injury, uninfected stage 3 and stage 4 pressure injury, and infected stage 3 and stage 4 pressure injury. Each scale is divided into three parts, including 1 item for hand hygiene, 6 items for material preparation, and 19 items for wound dressing change, for a total of 26 items. Medical staff or researchers will rate the participants' dressing change process as correctly performed, incorrectly performed, or not applicable, and the accuracy rate will be used as the evaluation result, that is, the total number of correctly performed questions minus the number of not applicable questions will be divided by the total number of the questions. The participants need to perform two actual dressing changes on the pressure injury, each time lasting approximately 15 minutes, totally approximately 30 minutes.

SECONDARY OUTCOMES:
Pressure injury dressing change of self-efficacy | 2 days
  This scale is designed to measure self-efficacy when changing the dressings of pressure injuries. It contains ten items and uses a four-point Likert scale with options ranging from "completely agree" to "completely disagree." The total score ranges from ten to forty, with a higher score indicating greater self-efficacy in dressing change for pressure injuries. Participants must fill out the scale twice, once before and after the intervention, each taking about 5 minutes, totally approximately 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: HSIAO-LING YANG, Ph. D., Study Chair — School of Nursing, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No